CLINICAL TRIAL: NCT01696786
Title: Oocyte Cryopreservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0903010292
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Fertility Preservation

ARMS (1):
- Oocyte cryopreservation (Experimental)
  Interventions: Procedure: Oocyte cryopreservation

INTERVENTIONS:
Procedure: Oocyte cryopreservation — Oocyte (egg) cryopreservation (freezing) to preserve fertility

SUMMARY:
The specific aim of this study is to further develop methods of oocyte cryopreservation and evaluate their impact on reproductive outcomes.

ELIGIBILITY:
Inclusion Criteria:

Any consenting female who wishes to freeze unfertilized oocytes and are:

1. at risk for ovarian hyperstimulation syndrome (enlarged ovaries with abdominal fluid accumulation) and postponement of pregnancy has been recommended.
2. a cancer patient anticipating treatment and have been cleared by the oncologists for ovarian stimulation.
3. a female who seeks to preserve her future fertility and does not wish to use donor or partner sperm to fertilize her eggs.
4. a donor egg recipient who elects to have some of the eggs obtained fertilized with husband/partner sperm and the rest cryopreserved for future use.
5. a patient for whom the partner's sperm retrieval or production has failed and donor sperm is not an option.
6. a patient who, for religious or ethical reasons, wants to limit the number of fresh oocytes exposed to sperm (fertilization) and do not want to either discard or donate the excess oocytes.

AND

1. has been clinically and psychologically approved for ovarian stimulation
2. age between 12 and 42 years, inclusive, at time of informed consent.
3. willing and able to comply with the protocol.
4. willing to provide follow-up information from her OB/GYN of any CVS/amniocentesis results, as well as information on obstetrical outcome.
5. agree to undergo intracytoplasmic sperm injection (ICSI) when oocytes are thawed.

For cancer patients:

1. No significant ovarian pathology as judged by physical exam and radiological studies;
2. Patient's general condition and prognosis deemed favorable for surgery and chemo/radio therapy;
3. No other major medical illness,
4. Oncologist approval for the ovarian stimulation and egg retrieval.

Exclusion Criteria:

Age > 42 Subjects who do not meet the inclusion criteria will be ineligible for participation in this study.

Max Age: 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-06 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Survival rate of cryopreserved oocytes with each cryopreservation method | 1 year
  Survival rate of cryopreserved oocytes with each cryopreservation method
Pregnancy rate following thawing/warming of oocytes | 1 year
  Pregnancy rate following thawing/warming of oocytes
Implantation rate per embryo transferred | 1 year
  Implantation rate per embryo transferred

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College, New York, New York, United States